CLINICAL TRIAL: NCT03438513
Title: Contribution of the Therapies of Resolution of Problem in the Care of the Natural Caregivers of Patients Affected by Neurodegenerative Disease Living at Home
Acronym: TRAMPD
Status: Withdrawn | Type: Observational
Why Stopped: Still no inclusion 10 months after the implementation visit. The study is outdated. Since, there has been "Alzheimer Plan" and establishment of external structures identical to the research project.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9727
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Neurodegenerative Diseases
Keywords: Caregivers; Burden; Coping; Quality of life; Problem solving therapy
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Problem Solving Therapy: This program is intended for caregivers to acquire techniques to manage stressful situations encountered in everyday life.
  Interventions: Behavioral: Problem Solving Therapy
- Speaking group: The group will be led by a psychologist.
  Interventions: Behavioral: Speaking group
- Standard medical care: Occupational Therapy Assessment Psychological assessment
  Interventions: Behavioral: Occupational Therapy Assessment; Behavioral: Psychological Assessment

INTERVENTIONS:
Behavioral: Occupational Therapy Assessment — The occupational therapy assessment includes a functional evaluation of the disorders impact (activities of daily living)
  Groups: Standard medical care
Behavioral: Psychological Assessment — It consists of a detailed history of the patient's experience, an evaluation with the patient (cognitive, emotional, motivational ...), an interview with the caregiver to see the repercussions of the disorders on a daily basis, how they are managed, and how they cope in order to give information and advice.
  Groups: Standard medical care
Behavioral: Problem Solving Therapy — Problem-solving learning program for all situations of daily living, done in groups (10 people per group)
  Groups: Problem Solving Therapy
Behavioral: Speaking group — Intervention, carried out in groups (10 people per group) which will consist of sharing experiences, sufferings, exchange and allow people who attend to share their experiences.
  Groups: Speaking group

SUMMARY:
The coverage of the caregivers of patients reached of neurodegenerative disease becomes essential. The psychic, physical but also social impacts for the caregivers are widely documented in the literature just like the stress associated with this role, we speak then about "burden of the caregivers". It seems that the caregivers set up little effective strategies of adaptation pulling fatal consequences on their well-being. He was shown in the literature, that a level of high stress is going to engender a decrease of mental flexibility and so entrainer a rigidity of adaptation.

To decrease the burden of the caregivers, numerous interventions were proposed. The analysis of the literature highlights that these interventions are rarely developed from theoretical models pulling(entailing) a stream of techniques proposed to the caregivers but without precise objective. The most effective interventions concerning the coverage(care) of the burden of the caregivers are the ones which are targeted and structured, those who put the helper in active position and who have an effect on the subjective burden. The cognitive-behavioral therapy (TCC) would seem particularly effective.

So, to modify the perception (collection) of the caregivers in front of cognitive, behavioral, functional modifications of their close friend(relation), to bring them to estimate positively their role and to favor the employment(use) of adaptive strategies turns out to be a privileged target of intervention to be used(employed) to improve the well-being of the caregivers and so decrease their burden.

Considering this, an intervention based on the techniques of resolution of problems (TRP) could show itself very relevant as specific coverage (care). The works concerning the contribution of the TRP and the adaptation generally concerning situations of health showed that this type(chap) of intervention facilitated an adapted situational coping, but also increased generally the social, academic and professional performances.

Various searches(researches) also showed that the resolution of problem is associated with indicators of adaptation at patients' nursing reached(affected) by Alzheimer's disease.

So we propose to the family caregivers a coverage(care) based on the therapy of resolution of problems taking support on the model of Lazarus's stress and Folkman and according to the model stemming from works of D' Zurilla and Nezu.

We make the hypothesis that this intervention is going to allow a decrease of the burden by allowing the caregivers to find a capacity to modulate their strategies to fit at best the evolutions of the clinical situation.

The main objective of our study is to compare the efficiency of a coverage(care) based on the Therapy of Resolution of Problems to a group of word and to that proposed at the moment within the pole of gerontology in the decrease of the burden of the caregivers of patients reached(affected) by neurodegenerative disease in 12 months. Our secondary objectives will concern the evolution of the burden in 6 months and the evolution of the strategies of coping, the anxious, depressive symptomatology, the quality of life, the mental flexibility in 6 and 12 months.

According to the data of the current literature, we expect a decrease of the psychological distress, an increase of the good(property) to be psychological. More specifically, by proposing an intervention targeted in particular at the management of the stress, the helper is going to acquire fitnesses which will have a long-lasting(sustainable) therapeutic effect.

By associating techniques of psychoeducation with techniques of management of the stress we hope we can propose a type(chap) of intervention suited to the natural caregivers to favor the preservation at home.

ELIGIBILITY:
Inclusion criteria:

- caregivers of patients affected by major neurocognitive disorder (cognitive decline which compromises the independence of the person). The symptoms vary according to the type of symptom, (Diagnostic and Statistical Manual 5) according to the definition of the European charter of the family helper " nobody not professional who helps main title partly or totally for one person dependent on its circle of acquaintances for the activities of the everyday life. This help can be lavished in a permanent way or not and can take various forms

Exclusion criteria:

* Diagnosis of major depression or other psychiatric affections
* Participation to another program of intervention (help to the caregivers, taken care TCC)
* Adults protected by the law
* Loss of liberty by court or administrative order.
* Absence of signature of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers of patients affected by major neurocognitive disorder
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
The evolution in 12 months of the burden of the caregivers estimated with the scale of burden of Zarit (ZBI) | 12 months after the inclusion
  Compare the efficiency of one taken care based on the therapy of resolution of problème